CLINICAL TRIAL: NCT06613386
Title: The Effects of an Information-Based Discharge Preparation Service on the Outcomes of Preterm Infant, Parent, and Hospital: a Randomized Controlled Trial
Brief Title: Effects of an Information-Based Discharge Service on Preterm Infants, Parents, and Hospitals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Chinese Medical Association (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: JSPH-NC-2022-18
Record Dates: First submitted 2024-08-27; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Patient Discharge; Infant, Premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: The study employs a prospective, double-arm, randomized controlled trial (RCT) design, conducted in the Neonatal Intensive Care Units (NICU) of a tertiary first-class hospital in Jiangsu Province, China.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IBDPS intervention (Experimental): Caregivers receive the IBDPS alongside usual care.
  * Grounded in the theories of empowerment and "Timing It Right" (TIR), the IBDPS delivers continuous, individualized support through an information-based platform from admission to one month postdischarge, facilitating seamless integration of discharge preparation across both online and offline environments.
  * Upon admission, caregivers register via WeChat, receiving tailored, stage-specific guidance on key topics such as "Growth," "Feeding," and "Sleep," aligned with the evolving needs of preterm infants. They can submit nursing concerns and assess their emotional state, with healthcare providers offering ongoing guidance. When the infant's condition stabilizes, caregivers can schedule NICU visits and engage in supervised bedside care training. Prior to discharge, hands-on training is provided. Postdischarge, caregivers upload growth data for continuous monitoring, with the option of home nurse visits.
  Interventions: Other: The information-based discharge preparation service (IBDPS)
- Usual care (No Intervention): Receive the usual care.
  * Routine admission education includes inpatient guidelines, breast milk storage, and receiving processes.
  * During hospitalization, healthcare providers are responsible for all infant care. Caregivers can visit three times a week at scheduled times, with visiting days arranged by the odd or even numbers of the inpatient ID. Visits are conducted via live video, allowing caregivers to consult with doctors about the infant's condition.
  * Upon discharge, healthcare providers educate caregivers on discharge precautions and preterm infant care methods.
  * Follow-up is conducted through phone calls and outpatient visits.

INTERVENTIONS:
Other: The information-based discharge preparation service (IBDPS) — The main modules of the IBDPS platform include:
  * Establishing information records for infants and parents.
  * Collaboratively identifying existing or potential caregiving challenges.
  * Assessing parents' emotional and psychological states, providing support and intervention.
  * Collaboratively establishing caregiving objectives with parents.
  * Collaboratively formulating and executing caregiving plans.
  * Assessing parental support resources, offering analysis, assistance, and necessary referrals.
  * Conducting outcome assessments.
  Arms: IBDPS intervention

SUMMARY:
Background:The Information-Based Discharge Preparation Service (IBDPS) supports parents of preterm infants during the transition from hospital to home, but its effectiveness has not been widely studied.

Objective:To evaluate the impact of IBDPS on parental readiness, caregiving skills, stress, satisfaction, infant development, readmission rates, length of stay, and hospital costs.

Design: A randomized controlled trial (RCT) in a NICU in Jiangsu Province, China.

Participants: Preterm infants and their parents.

Methods:Participants are randomly assigned to receive either IBDPS plus usual care (intervention group) or usual care alone (control group). Data on parental and infant outcomes are collected at various stages from admission to one month post-discharge, along with hospital metrics like length of stay and readmission rates.

DETAILED DESCRIPTION:
Participants are randomly allocated to the intervention and control groups. The intervention group receives the IBDPS in addition to the usual care, while the control group receives only the usual discharge education. The IBDPS, grounded in the theories of empowerment and "Timing It Right (TIR)," leverages an information-based platform to provide continuous, multidimensional, and customized support to parents from their infants' admission to one month post-discharge, ensuring seamless integration of discharge preparation both online and offline, and within and outside the hospital. Baseline data are collected at allocation (T1). Parental outcomes, including readiness for hospital discharge and stress, are assessed at T1, upon NICU entry (T2), and prior to discharge (T3), while caregiving skills are measured at T1, T2, T3, and one month post-discharge (T4). Parental satisfaction is measured at T3. Infant outcomes, such as weight, length, head circumference, breastfeeding rate, and feeding intolerance rate, are recorded at T1, T2, T3, and T4, with Neonatal Behavior Neurologic Assessment (NBNA) scores evaluated at T4. Hospital outcomes include length of stay and hospitalization costs, assessed at T3, and unplanned readmissions, recorded at T4.

ELIGIBILITY:
Inclusion Criteria for Infants:

* Infants with a gestational age of less than 37 weeks at birth.
* Written informed consent obtained from legal guardians.
* Neonates delivered at the study hospital or transferred within the first 24 hours of life.

Exclusion Criteria for Infants:

* Presence of major life-threatening congenital anomalies.
* Critical illness or conditions requiring immediate intensive intervention.
* Significant developmental abnormalities, including but not limited to severe congenital malformations, metabolic disorders, or central nervous system anomalies.

Removal Criteria for Infants:

* Infants who experience abnormal discharge due to treatment abandonment, death, or transfer to another facility.

Inclusion Criteria for Parents:

* Parents of infants born at less than 37 weeks of gestational age.
* Written informed consent provided by the parents.
* Ability to dedicate at least 4 hours per day to infant care.
* Adequate reading comprehension and proficiency in using electronic devices.
* If multiple caregivers are involved, the primary caregiver with the most hours of caregiving will be selected.

Exclusion Criteria for Parents:

* Health, familial, social, or language barriers that impair effective integration into the healthcare team.

Removal Criteria for Parents:

* Voluntary withdrawal from the study.
* Non-compliance with study protocols.

Max Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Readiness for Hospital Discharge Scale | From enrollment until the preterm infants discharge, with assessments at enrollment, parent entry into the NICU, and discharge,assessed up to 90 days.
  The Readiness for Hospital Discharge Scale (RHDS) - Parent Form was originally developed by Weiss et al. for assessing the readiness of parents for the discharge of their hospitalized children (0 to 18 years old). The Chinese version of the Readiness for Hospital Discharge Scale (C-RHDS) - Parent Form, adapted by Chen et al. with authorization from the original authors, is utilized to evaluate the readiness of parents for the discharge of preterm infants. This 22-item scale includes four dimensions: Knowledge (9 items), Physical-emotional Status (7 items), Pain Status (2 items), and Expected Support (4 items). Each item is scored on a scale from 0 to 10 (0 = worst; 10 = best), with total scores ranging from 0 to 220. Higher scores reflect better readiness for discharge. The overall Cronbach α coefficient for this scale is 0.91.

SECONDARY OUTCOMES:
Self-Assessment Questionnaire for Caregiving Ability of Parents of Preterm Infants | From enrollment until the preterm infants discharge, with assessments at enrollment, parent entry into the NICU, discharge,and one month after discharge,assessed up to 120 days.
  The Chinese version of the Self-Assessment Questionnaire for Caregiving Ability of Parents of Preterm Infants, developed by Meng et al., is used to evaluate the caregiving ability of parents with preterm infants. This questionnaire consists of 18 items rated on a Likert scale from 1 to 5 (1 = not at all familiar; 5 = very familiar). It is divided into three dimensions: Knowledge of Preterm Infant Care (7 items), Caregiving Skills (7 items), and Caregiving Ability (4 items). The total score ranges from 18 to 90, with higher scores indicating better caregiving ability. The Cronbach α coefficient for the overall scale is 0.956.

OTHER OUTCOMES:
Parental Stressor Scale: NICU | From the time of enrollment until the discharge of the preterm infant, with allocations made at enrollment, upon the parent entry into the NICU, and at discharge, assessed over a period of up to 90 days
  The Parental Stressor Scale: NICU (PSS: NICU) was originally developed by Miles and Funk et al. to measure parental stress during NICU hospitalization of their infants. The Chinese version of the Parental Stressor Scale: NICU (C-PSS: NICU), adapted by Li et al. with authorization from the original authors, uses a 5-point Likert scale (1 = no stress or anxiety; 5 = extreme stress or anxiety). This scale, consisting of 25 items, is divided into three dimensions: Infant Behavior and Appearance (13 items), Parental Role Alteration(7 items), and Sights and Sounds(5 items).The total score ranges from 25 to 125, with higher scores reflecting greater levels of parental stress and anxiety. The scale demonstrates strong internal consistency, with a Cronbach α coefficient of 0.856.
Parent Satisfaction Scale for Continuity of Care for Preterm Infants | Through the study completion, one month post-discharge,assessed up to 120 days.
  The Parent Satisfaction Scale for Continuity of Care for Preterm Infants, developed by Qian et al., can be used to assess parental satisfaction with discharge preparation services for preterm infants. This 21-item scale employs a 5-point Likert scale, where responses range from 0 (very dissatisfied) to 4 (very satisfied). The scale is structured into four dimensions: Nurse Appearance and Attitude(3 items),Continuity of Care Competence(11 items), Humanistic Quality(4 items), and Overall Evaluation of Continuity of Care Services(3 items).The scoring method is based on a percentage system, calculated as follows: (sum of scores for valid responses ÷ number of valid responses ÷ 4) × 100. Higher scores indicate greater satisfaction. The Cronbach α coefficient for the overall scale is 0.807.
Physical Development Outcomes | From enrollment until the preterm infants discharge, with assessments at enrollment, parent entry into the NICU, discharge,and one month after discharge,assessed up to 120 days.
  Indicators such as weight, length, and head circumference are measured using standardized neonatal techniques with calibrated scales and measuring tapes.
Neurobehavioral Development Outcomes | Through the study completion, one month post-discharge,assessed up to 120 days.
  Assessed using the Neonatal Behavior Neurologic Assessment (NBNA), a tool widely used in China to evaluate neurobehavioral development. NBNAis divided into five components: behavioral capability (6 items), passive muscle tone (4 items), active muscle tone (4 items), primitive reflexes (3 items), and general assessment (3 items). Each item is scored on a 3-point Likert scale ranging from 0 to 2, with a total possible score of 40. A score of ≤35 indicates abnormality.
Breastfeeding rate | From enrollment until the preterm infants discharge, with assessments at enrollment, parent entry into the NICU, discharge,and one month after discharge,assessed up to 120 days.
  The breastfeeding rate is calculated using the formula: (Number of breastfed infants ÷ Total number of infants) × 100%, recorded by nursing staff based on feeding logs.
Incidence of feeding intolerance | From enrollment until the preterm infants discharge, with assessments at enrollment, parent entry into the NICU, discharge,and one month after discharge,assessed up to 120 days.
  Incidence of feeding intolerance among preterm infants, as determined by the diagnostic criteria outlined in the first edition of Practical Neonatology, calculated using the formula: (Number of preterm infants identified with feeding intolerance ÷ Total number of preterm infants) × 100%, recorded by nursing staff based on feeding logs.
Length of Stay (LOS) | Until the discharge of the preterm infant, at the time of discharge,assessed up to 90 days.
  Length of Stay refers to the total duration of hospitalization for preterm infants during their initial NICU admission，collected the hospital Electronic Medical Record (EMR) system.
Hospitalization Costs | Until the discharge of the preterm infant,at the time of discharge,assessed up to 90 days.
  Hospitalization costs encompass the comprehensive financial expenditure associated with the NICU stay of preterm infants，collected from the hospital Electronic Medical Record (EMR) system
Readmission Rate Within One Month Post-Discharge | Through the study completion,one month post-discharge,assessed up to 120 days.
  The readmission rate within one month post-discharge refers to the proportion of preterm infants who required rehospitalization within 30 days following their discharge from the NICU, collected from the hospital Electronic Medical Record (EMR) system.

CONTACTS AND LOCATIONS:
Overall Officials: Caoyuan Wang, Master, Study Director — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang J, Cao M, Yue S, Yan J, Shang Y. Exploring Effect of Postdischarge Developmental Support Program on Preterm Infant Neurodevelopment and BDNF Gene DNA Methylation. Adv Neonatal Care. 2023 Apr 1;23(2):E50-E58. doi: 10.1097/ANC.0000000000001046. Epub 2022 Nov 21. PMID 36409665
- [Background] Cao G, Liu J, Liu M. Global, Regional, and National Incidence and Mortality of Neonatal Preterm Birth, 1990-2019. JAMA Pediatr. 2022 Aug 1;176(8):787-796. doi: 10.1001/jamapediatrics.2022.1622. PMID 35639401
- [Background] Smith VC, Mao W, McCormick MC. Changes in Assessment of and Satisfaction With Discharge Preparation From the Neonatal Intensive Care Unit. Adv Neonatal Care. 2021 Oct 1;21(5):E144-E151. doi: 10.1097/ANC.0000000000000862. PMID 33852448
- [Background] O'Connor M, Moriarty H, Schneider A, Dowdell EB, Bowles KH. Patients' and caregivers' perspectives in determining discharge readiness from home health. Geriatr Nurs. 2021 Jan-Feb;42(1):151-158. doi: 10.1016/j.gerinurse.2020.12.012. Epub 2021 Jan 11. PMID 33444923
- [Background] Hua W, Wang L, Li C, Simoni JM, Yuwen W, Jiang L. Understanding preparation for preterm infant discharge from parents' and healthcare providers' perspectives: Challenges and opportunities. J Adv Nurs. 2021 Mar;77(3):1379-1390. doi: 10.1111/jan.14676. Epub 2020 Nov 29. PMID 33249653
- [Background] Azzuqa A, Chuo J, Zenge J. Tele-medicine: Innovative tools for a safe transition to home in neonatal care. Semin Perinatol. 2021 Aug;45(5):151427. doi: 10.1016/j.semperi.2021.151427. Epub 2021 Apr 6. No abstract available. PMID 34006383
- [Background] Banerjee J, Aloysius A, Mitchell K, Silva I, Rallis D, Godambe SV, Deierl A. Improving infant outcomes through implementation of a family integrated care bundle including a parent supporting mobile application. Arch Dis Child Fetal Neonatal Ed. 2020 Mar;105(2):172-177. doi: 10.1136/archdischild-2018-316435. Epub 2019 Jun 21. PMID 31227521
- [Background] Richardson B, Dol J, Rutledge K, Monaghan J, Orovec A, Howie K, Boates T, Smit M, Campbell-Yeo M. Evaluation of Mobile Apps Targeted to Parents of Infants in the Neonatal Intensive Care Unit: Systematic App Review. JMIR Mhealth Uhealth. 2019 Apr 15;7(4):e11620. doi: 10.2196/11620. PMID 30985282
- [Background] Zhang R, Huang RW, Gao XR, Peng XM, Zhu LH, Rangasamy R, Latour JM. Involvement of Parents in the Care of Preterm Infants: A Pilot Study Evaluating a Family-Centered Care Intervention in a Chinese Neonatal ICU. Pediatr Crit Care Med. 2018 Aug;19(8):741-747. doi: 10.1097/PCC.0000000000001586. PMID 29781955
- [Background] Garfield CF, Lee YS, Kim HN, Rutsohn J, Kahn JY, Mustanski B, Mohr DC. Supporting Parents of Premature Infants Transitioning from the NICU to Home: A Pilot Randomized Control Trial of a Smartphone Application. Internet Interv. 2016 May;4(Pt 2):131-137. doi: 10.1016/j.invent.2016.05.004. Epub 2016 Jun 4. PMID 27990350